CLINICAL TRIAL: NCT02026778
Title: Comparison of the Effect of Ondansetron and Combined Ondansetron and Betahistine on Postoperative Nausea and Vomiting After Gynecological Laparoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 4-2013-0691
Record Dates: First submitted 2013-12-17; First posted 2014-01-03 (Estimated); Last update posted 2019-03-28 (Actual); Status verified 2015-05

CONDITIONS: Nausea and Vomiting
MeSH Terms: conditions — Nausea; Vomiting | interventions — Ondansetron

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ondansetron-betahistine (Experimental): ondansetron-betahistine group
  Interventions: Drug: ondansetron-betahistine
- ondansetron (Placebo Comparator): ondansetron group
  Interventions: Drug: ondansetron

INTERVENTIONS:
Drug: ondansetron — The ondansetron group is given placebo (pyridoxin) instead of betahistine.
  The ondansetron group is given ondansetron 4 mg bolus at the end of surgery and ondansetron 8 mg added to the IV-PCA.
  Arms: ondansetron
Drug: ondansetron-betahistine — The ondansetron-betahistine group is given betahistine 18mg orally in the morning of surgery and postoperative day 1.
  The ondansetron-betahistine group is given ondansetron 4 mg bolus at the end of surgery and ondansetron 8 mg added to the IV-PCA.
  Arms: ondansetron-betahistine

SUMMARY:
Many patients undergoing gynecologic laparoscopic surgery experience postoperative nausea and vomiting (PONV) despite prophylaxis and treatment with HT3 receptor antagonists such as ondansetron. Involvement of multiple types of receptors and factors may be a reason for inadequate control of PONV with a single agent. Betahistine, a histamine antagonist at H1 receptor and antagonist at H3 receptor, is widely used as a treatment of dizziness. Dizziness is one of the cause of nausea and vomiting. This study is to compare the effects of ondansetron and combined ondansetron and betahistine in preventing PONV in high-risk patients receiving intravenous opioid-based patient-controlled analgesia (IV-PCA) after gynecological laparoscopic surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patient scheduled for elective gynecological laparoscopic surgery
* American society of Anesthesiologists physical class I, Ⅱ, between the ages of 20 and 70 years

Exclusion Criteria:

* hepatorenal disease
* BMI > 35 kg/m2
* allergy to ondansetron or betahistine
* gastrointestinal disease
* vomiting within 24h
* administration of antiemetics or opioids within 24h
* QT prolongation (QTc > 440ms)
* Pheochromocytoma
* pregnant
* problem with communication

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2013-12; Primary Completion 2014-11-11 (Actual); Study Completion 2014-11-11 (Actual)

PRIMARY OUTCOMES:
postoperative nausea and vomiting | at postoperative 24h
  evaluation of nausea and vomiting with verbal rating scale (VRS, 0, no nausea; 10, worst imaginable nausea)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine, Yonsei University College of Medicine, Seoul, South Korea